CLINICAL TRIAL: NCT06334614
Title: iReach: a Novel Medical Device for Early Intervention for Visually Impaired Infants.
Brief Title: iReach: a Rehabilitative Medical Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Italiano di Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIT_iReach
Record Dates: First submitted 2024-03-20; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Blindness; Visual Impairment
Keywords: blindness; infants; rehabilitation; multisensory motor training; medical device
MeSH Terms: conditions — Blindness; Vision Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant masking because the clinical trial involves infants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iReach Device group (Experimental): The iReach Device group will undergo the clinical trial with the device in addition to the normal clinical activity
  Interventions: Device: iReach
- Normal clinical activity group (No Intervention): The Normal clinical activity group will continue their normal clinical activity

INTERVENTIONS:
Device: iReach — The iReach Device group will take part in playful multisensory motor and spatial activities for one month both at the clinic and at home with the medical device iReach.
  Arms: iReach Device group

SUMMARY:
The broad goal of this clinical trial is to demonstrate whether a one-month rehabilitative training with our medical device, iReach, can promote the recovery of spatial and sensorimotor abilities and the cortical reorganization process in children with visual impairment between 3 and 36 months of age.

DETAILED DESCRIPTION:
Development and clinical validation of a novel multisensory medical device: iReach. This device will be used for the rehabilitation and recovery of spatial and sensorimotor abilities compromised by early visual impairment (i.e., blindness or moderate to severe low vision) in children aged between 3 and 36 months. In addition to its clinical value, the investigators aim to fill a technological and methodological gap. Currently, there are no certified medical devices for early intervention, that is, systems that are intuitive, simple, and designed for rehabilitation in the early stages of development.

In detail, the goals of the current clinical trial are:

1. To verify that the number of adverse events is zero, considering reports from the attending physician;
2. To assess improvements in stationary and locomotion abilities, assessed with the Peabody Developmental Motor Scale (PDMS-2) indices;
3. To evaluate further improvements in i) reaction time (s) and frequency and accuracy of response (%) to uni- and multisensory (audio-tactile) stimulations; ii) time to reach and grasp an object (s); iii) number of attempts required to reach and grasp an object (%); iv) number of times the midline of the body is crossed to reach a lateral object (%); v) number of times an object is grasped with two hands if it is larger than the hand (%). These parameters will be extracted from video recordings;
4. To highlight changes in EEG power (dB) in the alpha band (8-12 Hz) measured in the occipital scalp area following rehabilitation with iReach.

iReach, is composed of two devices called Anchors, and a reference Tag, that can be placed either on both the body or external objects. Each Anchor measures its distance from the Tag and translates it into sensory feedback, whose intensity and time duration parameters are configurable. iReach can emit acoustic, vibrational, and RGB light stimuli, either alone or in combination, and is turned on via a button located on the external cover, which is manufactured through 3D printing.

This study is divided into two phases: usability and rehabilitation. The usability phase is aimed at defining the temporal durations of audio-tactile stimulations that will then be used in the rehabilitation phase. The patients enrolled in the iReach Device group of this phase will be involved in a one-month rehabilitation procedure (i.e., training) and will perform activities with iReach presented in the form of games that target localization, locomotion, grasping, and reaching skills. The training will be conducted both at home and at the clinical center and will be preceded and followed by two identical experimental sessions (pre- and post-training), which will monitor improvements in spatial and sensorimotor abilities following rehabilitation. Finally, an additional follow-up experimental session is planned four months after the post-training to verify whether these improvements are still present or not, both behaviorally and cortically. The participants enrolled in the Normal clinical activity group of the experimental phase will only be involved in the pre- and post-training sessions and the follow-up session without undergoing rehabilitation with iReach. The tasks the participants will have to undergo are designed for the specific age bin (i.e., 3-6 months, 6-12 months, 12-36 months)

ELIGIBILITY:
Inclusion Criteria:

* Obtaining Informed Consent;
* Age between 3 and 36 months;
* Normal vision or visual acuity between 0 and 4.7 cy/deg, assessed using the Teller Acuity Cards;
* Absence of concurrent therapies during the experimentation;
* Adequate cognitive ability for their age, assessed using the Reynell-Zinkin, Bayley III, and/or Griffiths scales;

Exclusion Criteria:

* Children with neurological disorders or cognitive delays (assessed using the Reynell-Zinkin, Bayley III, and/or Griffiths scales);
* Children affected by other sensory disabilities in addition to visual impairment (e.g., deafness) or with motor disorders;
* Premature infants with early gestational age (< 32 weeks);
* Children with diseases affecting the central nervous system or who have experienced epileptic seizures and/or convulsions in the six months before the start of the experimentation;
* Children with tactile hypersensitivity who are taking neuroactive drugs and substances or have taken them in the six months before the start of the experimentation;
* Children with auditory and/or peripheral motor disabilities;
* Children whose parents or legal guardians have not provided informed consent;

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Estimated)
Dates: Start 2024-12-08 (Estimated); Primary Completion 2025-05-08 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of Device Adverse Events | Month 1 - Month 12, the entire duration of the clinical trial
  Verification of the absence of device adverse events in the use of the medical device (MD);

SECONDARY OUTCOMES:
Change in motor skills after training with iReach medical device | Month 3 - Month 12
  The assessment of the change in certain motor skills (e.g., stability, and locomotion) after one month of intensive use of iReach. These changes will be quantified through the indices of the Peabody Developmental Motor Scales -2 (PDMS-2). The tasks included in these scales will be adapted to be executable by children with visual impairments. The PDMS-2 scales are widely used in clinical practice and allow for robust and reliable measurements. Higher scores result in better outcomes. The performance values are quantified through an indicator named "Total Motor Quotient," which spans from a minimum range equal to 35-69, representing a strong deficit, to a maximum range of 131-165, indicating the best performance.
Perceptual responses to multisensory stimuli | Month 1 - Month 12
  Evaluation of the number of correct responses and reaction times (in seconds), to uni- and multisensory (audio-tactile) stimuli.
Change in motor abilities following the rehabilitation with the iReach medical device | Month 1 - Month 12
  Evaluation of the changes in motor tasks in terms of: i) time to reach and grasp an object (in seconds) ii) number of attempts required to reach and grasp an object; iii) number of times the midline of the body is crossed to reach a lateral object; iv) number of times an object is grasped with two hands when its size exceeds that of the hand.
Variation in the power of the cortical activity following the rehabilitation with the iReach medical device | Month 1 - Month 12
  Evaluation of the variation in power expressed by the alpha band (8-12 Hz) of the EEG recorded in the occipital area (dB).

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Campus C, Signorini S, Vitali H, De Giorgis V, Papalia G, Morelli F, Gori M. Sensitive period for the plasticity of alpha activity in humans. Dev Cogn Neurosci. 2021 Jun;49:100965. doi: 10.1016/j.dcn.2021.100965. Epub 2021 May 21. PMID 34051686
- [Background] Cappagli G, Cocchi E, Gori M. Auditory and proprioceptive spatial impairments in blind children and adults. Dev Sci. 2017 May;20(3). doi: 10.1111/desc.12374. Epub 2015 Nov 27. PMID 26613827
- [Background] Cappagli G, Finocchietti S, Cocchi E, Giammari G, Zumiani R, Cuppone AV, Baud-Bovy G, Gori M. Audio motor training improves mobility and spatial cognition in visually impaired children. Sci Rep. 2019 Mar 1;9(1):3303. doi: 10.1038/s41598-019-39981-x. PMID 30824830
- [Background] Finocchietti S, Cappagli G, Ben Porquis L, Baud-Bovy G, Cocchi E, Gori M. Evaluation of the Audio Bracelet for Blind Interaction for improving mobility and spatial cognition in early blind children - A pilot study. Annu Int Conf IEEE Eng Med Biol Soc. 2015 Aug;2015:7998-8001. doi: 10.1109/EMBC.2015.7320248. PMID 26738148
- [Background] Gori M, Campus C, Signorini S, Rivara E, Bremner AJ. Multisensory spatial perception in visually impaired infants. Curr Biol. 2021 Nov 22;31(22):5093-5101.e5. doi: 10.1016/j.cub.2021.09.011. Epub 2021 Sep 22. PMID 34555348
- [Background] Setti W, Cuturi LF, Engel I, Picinali L, Gori M. The influence of early visual deprivation on audio-spatial working memory. Neuropsychology. 2022 Jan;36(1):55-63. doi: 10.1037/neu0000776. Epub 2021 Oct 14. PMID 34647755
- [Background] Vercillo T, Gori M. Attention to sound improves auditory reliability in audio-tactile spatial optimal integration. Front Integr Neurosci. 2015 May 7;9:34. doi: 10.3389/fnint.2015.00034. eCollection 2015. PMID 25999825
- See also: MySpace/iReach website — https://myspaceproject.eu/it/